CLINICAL TRIAL: NCT05366049
Title: The Effect of Injector and Pacifier Used in Oral Antipyretic Administration on the Vital Findings of the Child With Fever
Brief Title: The Effect of Methods Used in Oral Antipyretic Administration on the Vital Findings of the Child With Fever
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sermin Dİnç, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: E-59491012-604.01.02-2973
Record Dates: First submitted 2022-04-02; First posted 2022-05-09 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Fever; Heart Rate; Respiratory Rate; Pain
Keywords: children, oral medicine, medicine pacifier, injector, antipyretics
MeSH Terms: conditions — Fever; Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- using a medicine pacifier to give acetaminophen (Experimental)
  Interventions: Other: using a medicine pacifier to give acetaminophen
- using an enjector to give acetaminophen (Active Comparator)
  Interventions: Other: using a medicine pacifier to give acetaminophen

INTERVENTIONS:
Other: using a medicine pacifier to give acetaminophen — While giving acetaminophen, the effect on the amount of taking the drug, pain and vital parameters are observed by using the drug pacifier.

SUMMARY:
Fever, one of the most common clinical journeys of childhood, makes up a fraction of emergency room admissions. About us-30. High fever, which is one of the first schools in infancy and childhood, can cause health problems such as not applying or starting the intervention. The most preferred method in the fire; antipyretic drug treatment in the hospital is routine . Antipyretics play a role in control plans and estimations of facts for cars of cars, the importance of word of mouth has some problems. In children, hospital, health care, injectors are grown from the breeder after completion, they can be created by red supplementation from the effects such as rearing without completion . resistance children; aspiration is risky, wrong dose is administered. It is stated in relation to teachers and verbal medicines for health. Hansen et al. Working with 61 babies aged 0-24 months, using a pacifier injector and a normal injector, children and temperature monitors. They are from the nipple injector used by mothers and women. There is a need for a new modification in the existing oral drug applications that will be able to support the adaptation and readiness of the child and to be able to effectively administer the drug. This work; Two different methods used to give antipyretic (medication pacifier and colored injector) were planned to be performed as pain, fever and purpose of life (respiratory rate, planning CTA) for the child.

ELIGIBILITY:
Inclusion Criteria:

* Applying to the pediatric emergency department with a complaint of high fever (38ºC).
* Being prescribed an antipyretic (paracetamol) by a physician.
* Those whose parents are literate and agree to participate in the study.
* Patients with triage color classification Yellow and Green.
* Children between 0-24 months will be included in the study.

Exclusion Criteria:

* Having used antipyretics in the last 6 hours.
* Being prescribed an antipyretic other than paracetamol by the physician.
* Having trouble in sucking-swallowing coordination.
* Children with chronic disease and neuromotor developmental delay.

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Vital parameters | before oral medications
  Heart rate/minute

SECONDARY OUTCOMES:
Pain score | before oral medications
  Wong-baker pain scale. This scale is rated from 0 to 10. 0 is the pain of the pain, 10 is the pain to the beginning. shows. Pain by facial expression evaluation.

OTHER OUTCOMES:
vital parameters | before oral medications
  Respiratory rate/minute
vital parameters | before oral medications
  fever measurement (degrees centigrade)
Vital parameters | after medications 15 minute
  Heart rate/minute
Vital parameters | after medications 30 minute
  Heart rate/minute
Vital parameters | after medications 45 minute
  Heart rate/minute
Vital parameters | after medications 60 minute
  Heart rate/minute
Pain score | after medications 15 minute
  Wong-baker pain scale. This scale is rated from 0 to 10. 0 is the pain of the pain, 10 is the pain to the beginning. shows. Pain by facial expression evaluation.
Pain score | after medications 30 minute
  Wong-baker pain scale. This scale is rated from 0 to 10. 0 is the pain of the pain, 10 is the pain to the beginning. shows. Pain by facial expression evaluation.
Pain score | after medications 45 minute
  Wong-baker pain scale. This scale is rated from 0 to 10. 0 is the pain of the pain, 10 is the pain to the beginning. shows. Pain by facial expression evaluation.
Pain score | after medications 60 minute
  Wong-baker pain scale. This scale is rated from 0 to 10. 0 is the pain of the pain, 10 is the pain to the beginning. shows. Pain by facial expression evaluation.
vital parameters | after medications 15 minute
  Respiratory rate/minute
vital parameters | after medications 30 minute
  Respiratory rate/minute
vital parameters | after medications 45 minute
  Respiratory rate/minute
vital parameters | after medications 60 minute
  Respiratory rate/minute
vital parameters | after medications 15 minute
  fever measurement (degrees centigrade)
vital parameters | after medications 30 minute
  fever measurement (degrees centigrade)
vital parameters | after medications 45 minute
  fever measurement (degrees centigrade)
vital parameters | after medications 60 minute
  fever measurement (degrees centigrade)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Unisversity- Cerrahpasa, Istanbul, Fatih, Turkey (Türkiye)